CLINICAL TRIAL: NCT02220088
Title: The Efficacy and Safety of Retreatment With Transcatheter Arterial Infusion (TAI) for Patients Who Showed TACE-resistant: a Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Retreatment With TAI for Patients Who Showed TACE-resistant: a Randomized Controlled Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: protocol violation
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC201408
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; TACE; TACE failure; TACE refractoriness; TAI; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; Leucovorin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAI of FOLFOX (Experimental): Retreatment With Transcatheter arterial infusion of oxaliplatin , fluorouracil, and leucovorin
  Interventions: Procedure: TAI of FOLFOX
- Sorafenib (Active Comparator): treatment with sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Procedure: TAI of FOLFOX — Retreatment with TAI: administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: Transcatheter arterial infusion of oxaliplatin , fluorouracil, and leucovorin
  Arms: TAI of FOLFOX
Drug: Sorafenib — Accept sorafenib.
  Arms: Sorafenib

SUMMARY:
Transarterial chemoembolization (TACE) is considered the gold standard for treating intermediate-stage hepatocellular carcinoma (HCC). However, any treatment guidelines do not specify the criteria for repeating TACE. The study,conducted in Europe ，recently published in the journal of Hepatology shows the ART score of >=2.5 prior the second TACE identifies patients with a dismal prognosis who may not profit from further TACE sessions. However,in clinical practice，we also found some patients who showed TACE-resistant at the beginning of treatment may access to get objective response of retreatment with transcatheter arterial infusion (TAI). So the investigators conduct this prospective,randomized controlled study to find out whether the patient who showed TACE-resistant can obtain survival benefit from retreatment with TAI.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is considered the gold standard for treating intermediate-stage hepatocellular carcinoma (HCC). However, intermediate-stage HCC includes a heterogeneous population of patients with varying tumour burdens, liver function (Child-Pugh A or B) and disease aetiology.This suggests that not all patients with intermediate-stage HCC will derive similar benefit from transcatheter arterial infusion (TAI), and that some patients may benefit from other treatment options.

Repetition of TACE is based on evidence suggesting that one cycle of TACE may not be sufficient for effective treatment of intermediate-stage HCC and repeating TACE prolongs survival. However, intermediate-stage HCC patients often have unsatisfactory clinical outcomes with repeated TACE and there is not sufficiently addressed by existing guidelines include the criteria for repeating TACE and recommendations about the number of TACE cycles to be repeated before switching to another or no treatment.The study,recently published in the journal of Hepatology shows the ART score of >=2.5 prior the second TACE identifies patients with a dismal prognosis who may not profit from further TACE sessions.In clinical practice，however, we also found some patients who showed TACE-resistant at the beginning of treatment may access to get objective response of retreatment with TAI. So we conduct this prospective,randomized controlled study to find out whether the patient who showed TACE-resistant can obtain survival benefit from retreatment with TAI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients， > 18 years and <=70 years old diagnosed with HCC according to the European Association for the Study of the Liver (EASL) diagnostic criteria
* The patient has received 2 session of TACE
* TACE failure/refractoriness by Liver Cancer Study Group of Japan (LCSGJ) criteria
* Cirrhotic status of Child-Pugh class A
* The following laboratory parameters:

  * Platelet count ≥ 60,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Patients with complete response (CR) after the first TACE did not receive a further TACE session
* Eastern Cooperative Oncology Group (ECOG) >1
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Serious non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Severe Arterioportal Shunts or Arteriavein Shunts
* Known metastatic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 1 year

SECONDARY OUTCOMES:
Number of Adverse Events | 30 days
  All severe adverse events for the entire course of treatment
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Raoul JL, Sangro B, Forner A, Mazzaferro V, Piscaglia F, Bolondi L, Lencioni R. Evolving strategies for the management of intermediate-stage hepatocellular carcinoma: available evidence and expert opinion on the use of transarterial chemoembolization. Cancer Treat Rev. 2011 May;37(3):212-20. doi: 10.1016/j.ctrv.2010.07.006. Epub 2010 Aug 17. PMID 20724077
- [Result] Bolondi L, Burroughs A, Dufour JF, Galle PR, Mazzaferro V, Piscaglia F, Raoul JL, Sangro B. Heterogeneity of patients with intermediate (BCLC B) Hepatocellular Carcinoma: proposal for a subclassification to facilitate treatment decisions. Semin Liver Dis. 2012 Nov;32(4):348-59. doi: 10.1055/s-0032-1329906. Epub 2013 Feb 8. PMID 23397536
- [Result] Park JW, Amarapurkar D, Chao Y, Chen PJ, Geschwind JF, Goh KL, Han KH, Kudo M, Lee HC, Lee RC, Lesmana LA, Lim HY, Paik SW, Poon RT, Tan CK, Tanwandee T, Teng G, Cheng AL. Consensus recommendations and review by an International Expert Panel on Interventions in Hepatocellular Carcinoma (EPOIHCC). Liver Int. 2013 Mar;33(3):327-37. doi: 10.1111/liv.12083. Epub 2013 Jan 18. PMID 23331661
- [Result] Sieghart W, Hucke F, Pinter M, Graziadei I, Vogel W, Muller C, Heinzl H, Trauner M, Peck-Radosavljevic M. The ART of decision making: retreatment with transarterial chemoembolization in patients with hepatocellular carcinoma. Hepatology. 2013 Jun;57(6):2261-73. doi: 10.1002/hep.26256. Epub 2013 May 3. PMID 23316013
- [Result] Cheng AL, Amarapurkar D, Chao Y, Chen PJ, Geschwind JF, Goh KL, Han KH, Kudo M, Lee HC, Lee RC, Lesmana LA, Lim HY, Paik SW, Poon RT, Tan CK, Tanwandee T, Teng G, Park JW. Re-evaluating transarterial chemoembolization for the treatment of hepatocellular carcinoma: Consensus recommendations and review by an International Expert Panel. Liver Int. 2014 Feb;34(2):174-83. doi: 10.1111/liv.12314. Epub 2013 Nov 20. PMID 24251922
- [Result] Hucke F, Sieghart W, Pinter M, Graziadei I, Vogel W, Muller C, Heinzl H, Waneck F, Trauner M, Peck-Radosavljevic M. The ART-strategy: sequential assessment of the ART score predicts outcome of patients with hepatocellular carcinoma re-treated with TACE. J Hepatol. 2014 Jan;60(1):118-26. doi: 10.1016/j.jhep.2013.08.022. Epub 2013 Sep 3. PMID 24012941
- [Result] Yousuf F, Cross TJ, Palmer D. The ART strategy: sequential assessment of the ART score predicts outcome of patients with hepatocellular carcinoma re-treated with TACE. J Hepatol. 2014 Jul;61(1):175. doi: 10.1016/j.jhep.2014.02.032. Epub 2014 Mar 18. No abstract available. PMID 24657396